CLINICAL TRIAL: NCT03184220
Title: Treatment of Cervical Syndrome With Myofascial Therapies
Acronym: MRH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, Clinical Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32/16
Record Dates: First submitted 2017-05-18; First posted 2017-06-12 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Cervical Syndrome
Keywords: Neck Pain; Physical Therapy Modalities; Fascia; Manual Therapy; Massage
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CLINICAL TRIAL WITH BLIND EVALUATION BY THIRD PARTIES, LONGITUDINAL AND PROSPECTIVE.
Who Masked: Investigator
Masking Description: Blind researcher
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Patients who are pregnant, have pacemaker and those surgically operated cervical spine patients who have been treated with myofascial therapy a month earlier.
  Multimodal physical therapy program includes:
  Myofascial syndrome cervical therapy treatment.
  Interventions: Procedure: Physiotherapy treatment
- CONTROL GROUP (Experimental): Multimodal physical therapy program includes:
  * ultrasound therapy (US),
  * transcutaneous electric nerve stimulation (TENS)
  * massage.
  Interventions: Procedure: Physiotherapy treatment

INTERVENTIONS:
Procedure: Physiotherapy treatment — The MRT group was treated five times with several maneuvers. Each maneuver was performed once per session by slow and progressive application of a light force. The whole procedure lasted no more than 45 minutes. The treatment included four basic maneuvers.
  * Suboccipital induction
  * Posterior elongation of the cervical fascia in Supine position
  * Assisted cervical fascia
  * Myofascial induction of sternocleidomastoid
  Arms: EXPERIMENTAL GROUP
Procedure: Physiotherapy treatment — The PT group will treated during two weeks (ten days/week) with ultrasound therapy (US), transcutaneous electric nerve stimulation (TENS) and massage, in this order. Ultrasound will applied in pulse mode at an intensity of 1 megahertz for 10 minutes in the sub-occipital region and the vicinity of the trapezius muscles. TENS will applied with a pulse duration of 250 microseconds at a frequency of 80 Hertz for 20 minutes in the sub-occipital region and the trapezoids. Deep massage was applied at a slow speed for 20 minutes using sliding neutral creams. Massage therapy included gliding and kneading techniques applied over trapezius (upper, lower and middle fibers), splenius capitis and levator scapulae muscles with a therapeutic intention.
  Arms: CONTROL GROUP

SUMMARY:
This study aimed to investigate the effects of myofascial release therapy (MRT) for improving pressure pain thresholds (PPTs), range of motion and pain in patients with mechanical neck pain (NP).

DETAILED DESCRIPTION:
Fifty-four participants with NP were randomly allocated to either an MRT (five sessions) or a physical therapy (PT) groups (ten sessions) during two weeks. Multimodal PT program included: ultrasound therapy (US), transcutaneous electric nerve stimulation (TENS) and massage. Visual Analogue Scale (VAS), range of motion and (CROM) PPTs in sub-occipital and upper trapezius muscles were measured at baseline, at the end of treatment and at 1 month follow-up. T-tests and a repeated-measures multivariate analysis of variance (RM-MANOVA) were used for VAS, CROM and PPTs, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged between 20 and 60 years, in an active state of pain and diagnosed with muscle breakdown

Exclusion Criteria:

- Patients who are pregnant, have pacemakers and surgically operated in the area to be treated

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
The intensity of cervical pain | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.

SECONDARY OUTCOMES:
The intensity of cervical pain | Four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.
The intensity of cervical pain | Eight weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of cervical pain, and the worst and lowest level of pain experienced in the preceding week in the cervical area.
Active cervical range of motion | Baseline, four weeks and eight weeks
  Measured by goniometer type crom
Pressure pain thresholds in cervical trigger points | Baseline, four weeks and eight weeks
  Pressure pain thresholds (PPTs) will be measured with a pressure algometer (Baseline, Pain TestTM, Wagner Instruments). The clinimetric properties of this instrument have been evaluated previously. The PPT will the point at which pressure elicited pain and will presented as kilograms per square centimeter. All measurements will be conducted by the same well-trained physician.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodriguez Huguet, Principal Investigator — University of Cadiz
Locations (1):
- Policlínica Santa maría, Cadiz, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Leaver AM, Maher CG, McAuley JH, Jull G, Latimer J, Refshauge KM. People seeking treatment for a new episode of neck pain typically have rapid improvement in symptoms: an observational study. J Physiother. 2013 Mar;59(1):31-7. doi: 10.1016/S1836-9553(13)70144-9. PMID 23419913
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Palmlof L, Skillgate E, Alfredsson L, Vingard E, Magnusson C, Lundberg M, Holm LW. Does income matter for troublesome neck pain? A population-based study on risk and prognosis. J Epidemiol Community Health. 2012 Nov;66(11):1063-70. doi: 10.1136/jech-2011-200783. Epub 2012 Mar 12. PMID 22412154
- [Background] Noormohammadpour P, Mansournia MA, Koohpayehzadeh J, Asgari F, Rostami M, Rafei A, Kordi R. Prevalence of Chronic Neck Pain, Low Back Pain, and Knee Pain and Their Related Factors in Community-Dwelling Adults in Iran: A Population-based National Study. Clin J Pain. 2017 Feb;33(2):181-187. doi: 10.1097/AJP.0000000000000396. PMID 27258995
- [Background] De Pauw R, Coppieters I, Kregel J, De Meulemeester K, Danneels L, Cagnie B. Does muscle morphology change in chronic neck pain patients? - A systematic review. Man Ther. 2016 Apr;22:42-9. doi: 10.1016/j.math.2015.11.006. Epub 2015 Dec 11. PMID 26724855
- [Background] Rodriguez-Fuentes I, De Toro FJ, Rodriguez-Fuentes G, de Oliveira IM, Meijide-Failde R, Fuentes-Boquete IM. Myofascial Release Therapy in the Treatment of Occupational Mechanical Neck Pain: A Randomized Parallel Group Study. Am J Phys Med Rehabil. 2016 Jul;95(7):507-15. doi: 10.1097/PHM.0000000000000425. PMID 26745225
- [Background] Tozzi P, Bongiorno D, Vitturini C. Fascial release effects on patients with non-specific cervical or lumbar pain. J Bodyw Mov Ther. 2011 Oct;15(4):405-16. doi: 10.1016/j.jbmt.2010.11.003. Epub 2011 Jan 8. PMID 21943614
- [Background] Lluch E, Nijs J, De Kooning M, Van Dyck D, Vanderstraeten R, Struyf F, Roussel NA. Prevalence, Incidence, Localization, and Pathophysiology of Myofascial Trigger Points in Patients With Spinal Pain: A Systematic Literature Review. J Manipulative Physiol Ther. 2015 Oct;38(8):587-600. doi: 10.1016/j.jmpt.2015.08.004. Epub 2015 Sep 19. PMID 26387860
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Munoz-Munoz S, Munoz-Garcia MT, Alburquerque-Sendin F, Arroyo-Morales M, Fernandez-de-las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in individuals with mechanical neck pain. J Manipulative Physiol Ther. 2012 Oct;35(8):608-13. doi: 10.1016/j.jmpt.2012.09.003. PMID 23158466
- [Background] Jeon JH, Jung YJ, Lee JY, Choi JS, Mun JH, Park WY, Seo CH, Jang KU. The effect of extracorporeal shock wave therapy on myofascial pain syndrome. Ann Rehabil Med. 2012 Oct;36(5):665-74. doi: 10.5535/arm.2012.36.5.665. Epub 2012 Oct 31. PMID 23185731
- [Background] Cook AJ, Wellman RD, Cherkin DC, Kahn JR, Sherman KJ. Randomized clinical trial assessing whether additional massage treatments for chronic neck pain improve 12- and 26-week outcomes. Spine J. 2015 Oct 1;15(10):2206-15. doi: 10.1016/j.spinee.2015.06.049. Epub 2015 Jun 19. PMID 26096474
- [Background] Lopez-Lopez A, Alonso Perez JL, Gonzalez Gutierez JL, La Touche R, Lerma Lara S, Izquierdo H, Fernandez-Carnero J. Mobilization versus manipulations versus sustain apophyseal natural glide techniques and interaction with psychological factors for patients with chronic neck pain: randomized controlled trial. Eur J Phys Rehabil Med. 2015 Apr;51(2):121-32. Epub 2014 Oct 9. PMID 25296741
- [Background] Liptan G, Mist S, Wright C, Arzt A, Jones KD. A pilot study of myofascial release therapy compared to Swedish massage in fibromyalgia. J Bodyw Mov Ther. 2013 Jul;17(3):365-70. doi: 10.1016/j.jbmt.2012.11.010. Epub 2013 Jan 3. PMID 23768283
- [Background] Moraska AF, Stenerson L, Butryn N, Krutsch JP, Schmiege SJ, Mann JD. Myofascial trigger point-focused head and neck massage for recurrent tension-type headache: a randomized, placebo-controlled clinical trial. Clin J Pain. 2015 Feb;31(2):159-68. doi: 10.1097/AJP.0000000000000091. PMID 25329141
- [Background] Saiz-Llamosas JR, Fernandez-Perez AM, Fajardo-Rodriguez MF, Pilat A, Valenza-Demet G, Fernandez-de-Las-Penas C. Changes in neck mobility and pressure pain threshold levels following a cervical myofascial induction technique in pain-free healthy subjects. J Manipulative Physiol Ther. 2009 Jun;32(5):352-7. doi: 10.1016/j.jmpt.2009.04.009. PMID 19539117
- [Background] Yuan SL, Matsutani LA, Marques AP. Effectiveness of different styles of massage therapy in fibromyalgia: a systematic review and meta-analysis. Man Ther. 2015 Apr;20(2):257-64. doi: 10.1016/j.math.2014.09.003. Epub 2014 Oct 5. PMID 25457196
- [Background] Calixtre LB, Moreira RF, Franchini GH, Alburquerque-Sendin F, Oliveira AB. Manual therapy for the management of pain and limited range of motion in subjects with signs and symptoms of temporomandibular disorder: a systematic review of randomised controlled trials. J Oral Rehabil. 2015 Nov;42(11):847-61. doi: 10.1111/joor.12321. Epub 2015 Jun 7. PMID 26059857
- [Background] Serrano-Aguilar P, Kovacs FM, Cabrera-Hernandez JM, Ramos-Goni JM, Garcia-Perez L. Avoidable costs of physical treatments for chronic back, neck and shoulder pain within the Spanish National Health Service: a cross-sectional study. BMC Musculoskelet Disord. 2011 Dec 21;12:287. doi: 10.1186/1471-2474-12-287. PMID 22188790
- [Background] Wong JJ, Shearer HM, Mior S, Jacobs C, Cote P, Randhawa K, Yu H, Southerst D, Varatharajan S, Sutton D, van der Velde G, Carroll LJ, Ameis A, Ammendolia C, Brison R, Nordin M, Stupar M, Taylor-Vaisey A. Are manual therapies, passive physical modalities, or acupuncture effective for the management of patients with whiplash-associated disorders or neck pain and associated disorders? An update of the Bone and Joint Decade Task Force on Neck Pain and Its Associated Disorders by the OPTIMa collaboration. Spine J. 2016 Dec;16(12):1598-1630. doi: 10.1016/j.spinee.2015.08.024. Epub 2015 Dec 17. PMID 26707074
- [Background] Cagnie B, Castelein B, Pollie F, Steelant L, Verhoeyen H, Cools A. Evidence for the Use of Ischemic Compression and Dry Needling in the Management of Trigger Points of the Upper Trapezius in Patients with Neck Pain: A Systematic Review. Am J Phys Med Rehabil. 2015 Jul;94(7):573-83. doi: 10.1097/PHM.0000000000000266. PMID 25768071
- [Background] Bervoets DC, Luijsterburg PA, Alessie JJ, Buijs MJ, Verhagen AP. Massage therapy has short-term benefits for people with common musculoskeletal disorders compared to no treatment: a systematic review. J Physiother. 2015 Jul;61(3):106-16. doi: 10.1016/j.jphys.2015.05.018. Epub 2015 Jun 17. PMID 26093806
- [Background] Fletcher JP, Bandy WD. Intrarater reliability of CROM measurement of cervical spine active range of motion in persons with and without neck pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):640-5. doi: 10.2519/jospt.2008.2680. PMID 18827326